CLINICAL TRIAL: NCT05831995
Title: A Phase I, First-In-Human, Multicenter, Open Label, Dose Escalation and Dose Expansion Study to Evaluate the Safety and Efficacy of ABM-168 Administered Orally in Adult Patients with Advanced Solid Tumors
Brief Title: Safety and Effectiveness of ABM-168 in Adults with Advanced Solid Tumors.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to development strategy change.
Sponsor: ABM Therapeutics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ABM168X1101
Record Dates: First submitted 2023-03-07; First posted 2023-04-27 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Advanced Solid Tumor; RAS Mutation; RAF Mutation; NF1 Mutation
Keywords: Melanoma; Glioblastoma; Colorectal cancer; Lung cancer; Pancreatic cancer; Metastatic brain tumors; Primary CNS tumors; All Solid Tumors
MeSH Terms: conditions — Melanoma; Glioblastoma; Colorectal Neoplasms; Lung Neoplasms; Pancreatic Neoplasms; Brain Neoplasms

STUDY DESIGN:
Intervention Model Description: Study consists of two parts:
  * Part A: ABM-168 Dose Escalation and DLT Dose Confirmation
  * Part B: Dose Expansion (ABM-168 Monotherapy)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Experimental Monotherapy Dose Escalation (Experimental): A classic "3+3" design will be used to explore the maximum tolerated dose (MTD) and to determine the recommended phase II dose (RP2D). Three to four patients will be enrolled to ensure at least 3 evaluable patients for DLT (Dose Limiting Toxicity). ABM-168 monotherapy will be conducted in seven provisional dose levels starting at 0.5mg oral administration per day and up to and including 12mg oral administration. Each treatment cycle is 28-days. DLT will be evaluated in the first 28-day cycle. Patients will receive daily doses of ABM-168 until disease progression; intolerable toxicity; withdrawal consent; or other clinical observation is met.
  Interventions: Drug: ABM-168
- Experimental Monotherapy Dose Expansion-1 (Experimental): Expansion will be conducted in the adult patients with advanced solid tumors that carry either RAS, RAF or NF-1 mutations. Cohort EX1 will enroll the patients with preferred indications (i.e., melanoma, colon cancer, lung cancer, and pancreatic carcinoma) who had confirmed RAS, RAF or NF-1 mutations and measurable target lesion(s) at baseline. Patients with measurable brain metastases lesion(s) at baseline are highly preferred. Up to 15 evaluable patients will be enrolled for each into each preferred indication. Other indication(s) that show confirmed response, complete response (CR) or partial response (PR) in at least one subject in the dose escalation study will facilitate the preferred indication(s) for Cohort EX1 enrollment as well.
  Interventions: Drug: ABM-168
- Experimental Monotherapy Dose Expansion-2 (Experimental): Expansion will be conducted in the adult patients with advanced solid tumors that carry either RAS, RAF or NF-1 mutations. Cohort EX2 will enroll the patients who had primary CNS tumors with confirmed RAS, RAF or NF-1 mutations at baseline. Up to 30 evaluable patients will be enrolled.
  Interventions: Drug: ABM-168

INTERVENTIONS:
Drug: ABM-168 — Dosage: 0.5 mg; 2 mg; 6 mg; once daily by oral administration

SUMMARY:
This is a Phase 1, First-in-Human (FIH), open-label, multicenter, dose escalation and dose expansion study to evaluate the safety, tolerability, pharmacokinetics and preliminary anti-tumor activity of ABM-168 in adult patients with RAS or RAF or NF-1 mutated advanced solid tumors as ABM-168 may have a significant effect in inhibiting cell growth.

DETAILED DESCRIPTION:
This is a First-in-Human (FIH), open-label, multicenter, dose escalation and dose expansion, Phase I study of ABM-168, for the treatment of advanced solid tumors in adult patients.

The study consists of two parts:

Part A: Dose escalation. The starting dose of ABM-168 is 0.5 mq po qd, and dose escalation will be guided by a "3+3" design. ABM-168 will be administered once daily on a continuous schedule. Each treatment cycle consists of 28 days.

Part B: Dose Expansion. Expansion will be conducted in the adult patients with advanced solid tumors that carry either RAS, RAF or NF-1 mutations. There are two cohorts for Dose Expansion: Patients will be enrolled into either Dose Expansion Cohort 1 (EX1) or Dose Expansion Cohort 2 (EX2).

* Cohort EX1: Patients enrolled will have preferred indications (i.e., melanoma, colon cancer, lung cancer, and pancreatic carcinoma) who had confirmed RAS, RAF or NF-1 mutations and measurable lesion(s) at the beginning of the study. Patients with measurable brain lesions(s) which have metastasized are highly preferred.
* Cohort EX2: Patients enrolled will have primary CNS (Central Nervous System tumors with confirmed RAS, RAF or NF-1 mutations.

Dose limiting toxicity (DLT) will be evaluated and managed per the pre-defined DLT criteria and rules specified in the protocol. MTD (Maximum Tolerated Dose) and/or RP2D will be determined based on the totality of safety, clinical pharmacokinetics, and efficacy data from all evaluable patients enrolled and in treated in both dose escalation cohorts and dose expansion cohorts. The RP2D (recommended phase II dose) could be the MTD, or alternatively a dose recommended by the SMC (Safety Monitoring Committee) if no MTD is determined in the dose escalation and/or dose expansion.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects age 18 years and older who are able to sign informed consent and comply with the protocol
2. Patients with histologically or cytologically documented, locally advanced, or metastatic solid tumor malignancy that has either:

   1. failed prior standard therapy; or
   2. exhausted all existing standard therapy; or
   3. standard therapy is not considered appropriate per subject and/or investigator. No limitation on the lines of previous standard therapy received.
3. Patients with asymptomatic or symptomatic but stable brain metastases or CNS primary malignancies who meet following criteria specifically:

   * Asymptomatic, brain metastases or primary CNS tumors;
   * Stable symptomatic brain metastases or CNS primary tumors not requiring steroids treatment or receiving steroids treatment (dexamethasone or equivalent) with total daily dosage no more than 4 mg, with a stable or reduced dosage of steroids within 2 weeks prior to the planned first dose
4. ECOG performance score of 0 or 1, or Karnofsky performance score of ≥ 70.
5. ≥ 3 months life expectancy
6. Receiving no blood transfusions or granulocyte colony-stimulating factor (G-CSF) or other hematopoietic stimulating factors within 2 weeks prior to the planned first dosing. Adequate organ function confirmed at screening as evidenced by:

   * Absolute Neutrophil Count (ANC) ≥ 1.5 × 10^9/L
   * Hemoglobin (Hgb) ≥ 90 g/dL
   * Platelets (Plt) ≥ 75 ×10^9/L
   * AST/ALT ≤ 2.5 × Upper Limit of Normal (ULN) or ≤ 5.0 × ULN if liver metastases are present
   * Total bilirubin ≤ 1.5 × ULN, or direct bilirubin < ULN (for patients with total bilirubin levels >1.5 ×ULN)
   * Calculated creatinine clearance ≥ 60 mL/min
   * International normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN, if received no anti-coagulation medication(s); INR ) ≤ ULN, if received anti-coagulation medication(s).
   * Average QTcF ≤ 470 ms per Fridericia formula
7. Negative Hepatitis B Surface Antigen (HBsAg) at screening, or positive HBsAg with HBV DNA below LLN.

   Notes: Manage HBsAg positive subject according to the institutional standard practices (i.e., monitor HBV DNA, prescribe anti-HBV therapy as needed, etc.)
8. Hepatitis C Virus (HCV) viral load below limit of quantification at screening, or positive HCV antibody with negative HCV-RNA.

   Notes: Only conduct HCV antibody and/or HCV-RNA assay in the subjects with prior history of HCV infection.
9. Negative HIV at screening, or patients with prior history of HIV infection, CD4+ T-cell (CD4+) counts ≥ 350 cells/μL and without a history of AIDS-defining opportunistic infections.
10. Negative serum pregnancy test within 72 hours before starting study treatment in all pre-menopausal women and women < 12 months after the onset of menopause
11. Must agree to take sufficient contraceptive methods to avoid pregnancy, starting from the consent until 3 months post receiving the last dose of study drug
12. Able to swallow capsule as a whole
13. [Dose Escalation Cohorts Only] Subject with evaluable but not measurable lesion is allowed for enrollment.
14. [Dose Expansion Cohorts Only] Subject must have at least one measurable lesion, intracranial or extracranial, detected at the baseline assessment by RECIST V1.1 criteria for solid tumors or the RANO criteria for primary CNS tumors, such as gliomas.

    * The lesion(s) exposed to previous radiation cannot be selected as target lesion(s) at baseline assessment, unless obvious progression of the lesion(s) can be proved via the imaging assessment;
    * For solid tumor brain metastases lesions:
    * If the longest diameter of the measurable intracranial lesion is < 0.5 cm, then at least one extracranial measurable lesion should exist [Dose Expansion cohorts only];
    * Measurable brain lesions that are 0.5 - 3 cm in longest diameter as defined by the modified RECIST V1.1 criteria are allowed.
    * Brain lesion size > 3 cm is not eligible

Exclusion Criteria:

1. Women who are pregnant or breast-feeding.
2. Have leptomeningeal disease (LMD).
3. Have a history of stroke within 6 months prior to the first dose.
4. Have impaired cardiac function or clinically significant cardiovascular disease(s) including but not limited to any of the following:

   * Left ventricular ejection fraction (LVEF) < 50% as determined by cardiac ultrasound.
   * Congenital long QT syndrome.
   * Grade 2 type II AV block or grade 3 AV block.
   * Unstable angina within 6 months prior to the first dose.
   * Acute myocardial infarction within 6 months prior to the first dose.
   * ≥ Class III heart failure per New York Heart Association (NYHA) functional classification within 6 months prior to the first dose.
   * ≥ CTCAE Grade 2 ventricular arrhythmia within 6 months prior to study initiation.
5. Have uncontrolled hypertension at screening, with systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg after receiving anti-hypertension treatment.
6. Have unresolved ≥ CTCAE Grade 2 diarrhea at the time of the first dose; or have gastrointestinal impairment conditions or diseases that significantly alter ABM-168 absorption at screening per investigator (e.g., ulcerative disease, poorly controlled nausea, vomiting, malabsorption syndrome, or small intestine dissection)
7. Have ≥ CTCAE Grade 2 eye diseases at screening, such as conjunctival mixed cellular inflammation, corneal ulcer.
8. Have severe chronic or active infection requiring intravenous antibiotic treatment(s) within 2 weeks prior to the first dose, including but not limited to hospitalization due to infection complications, bacteremia, severe pneumonia or active tuberculosis.

   Notes:
   * Subjects with topical fungal infection of the skin or nails are eligible for study enrollment.
   * Subjects receiving prophylactic antibiotics (e.g., to prevent urinary tract infections or exacerbations of chronic obstructive pulmonary disease), except for the antibiotics prohibited per protocol, are eligible for study enrollment.
9. Received solid organ or hematopoietic bone marrow/stem cell transplantation within 5 years prior to the screening.
10. Received chemotherapy, targeted therapy or immunotherapy within 4 weeks prior to the first dose, except for fluorouracil or small molecule target therapy.

    Notes: Fluorouracil or small molecule target therapy received within five half-life or 2 weeks (whichever is longer) prior to the first dose is not allowed.
11. Received anti-tumor Chinese herbal medicines or proprietary Chinese medicines within 2 weeks prior to the first dose.
12. Received extensive prior radiotherapy to more than 30% of bone marrow reserves; or received Whole Brain Radiation Therapy (WBRT) within 4 weeks prior to the first dose; or received palliative radiotherapy for non-target lesions (e.g., bone radiotherapy for pain relief), including stereotactic body radiotherapy (SBRT) and stereotactic radiosurgery (SRS) within 2 weeks prior to the first dose.
13. Have adverse reactions related to previous anti-tumor therapy that have not recovered to ≤ CTCAE Grade 1 or previous baseline at screening.

    Notes: Subjects with alopecia, or ≤ CTCAE Grade 2 peripheral neuropathy, or hypothyroidism stabilized by hormone replacement therapy, etc. are allowed for the enrollment.
14. Have undergone major surgery within 4 weeks prior to the first dose, or have not recovered from the side effects of major surgery, or expect to receive major surgery during study treatment.

    Notes: For subject who has recovered from major surgery per investigator, a minimum of 2 weeks washout between the major surgery and the first dose is required.
15. Received therapeutic doses of warfarin sodium or any other coumarin derivative anticoagulant at screening.
16. Received systemic corticosteroids within 2 weeks prior to the first dose, or not recovered from adverse effects of previous corticosteroids treatment, except those as described in the inclusion criteria for subjects with brain metastases.

    Notes: Subjects who received topical, intranasal or inhaled glucocorticoids; or subjects who received physiologic dose of steroids for adrenal replacement; subjects who received single-use glucocorticoids for the prevention of contrast medium allergy prior to the imaging enhancement examinations are eligible for study enrollment.
17. Have history of alcohol abuse or alcohol addiction within 3 months prior to the first dose.
18. Have known, documented, or suspected history of substance abuse, except for opioids etc. prescribed for pain relief.
19. Have past or current evidence of conditions that may affect the study results per investigator, or any conditions, treatment or laboratory abnormalities that may interfere with the subject's participation in the trial and study compliance.
20. Other severe and/or poorly controlled concomitant diseases that may cause unacceptable safety risks or affect compliance with the study protocol.
21. History of immunodeficiency, including a positive HIV antibody test.
22. Other circumstances deemed as not suitable for study enrollment per investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Determine Dose Limiting Toxicity (DLT) and/or Recommended Phase 2 dose (RP2D) | Day 28 after last dosing.
  Dose limiting toxicities (DLT) which defines the MTD/RP2D
Safety and tolerability-Incident Rate. | Day 28 after last dosing.
  Safety and tolerability of ABM-168 monotherapy as determined by incident rate.
Safety and tolerability, severity per Common Toxicity Criteria for Adverse Events (CTCAE v5.0) | Day 28 after last dosing.
  Safety and tolerability of ABM-168 monotherapy as determined by severity. Adverse events will be assessed according to the National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE) version 5.0. For consistency, Version 5.0 will be used throughout the trial regardless of any subsequent versions of the CTCAE criteria that may become available. If CTCAE grading does not exist for a specific adverse event, the severity should be assessed based on the general guidelines outlined in CTCAE v5.0.
Safety and tolerability-AE causality. | Day 28 after last dosing.
  Safety and tolerability of ABM-168 monotherapy as determined by causality of adverse events (AEs).
Safety and tolerability-Lab abnormalities. | Day 28 after last dosing.
  Safety and tolerability of ABM-168 monotherapy as determined by clinically significant abnormalities in clinical laboratory testing.
Safety and tolerability-Body Temperature. | Day 28 after last dosing.
  Safety and tolerability of ABM-168 monotherapy as determined by body temperature changes from base-line in Fahrenheit.
Safety and tolerability-Heart Rate | Day 28 after last dosing.
  Safety and tolerability of ABM-168 monotherapy as determined by heart rate changes from base-line in BPM (beats per minute).
Safety and tolerability-Pulse Rate | Day 28 after last dosing.
  Safety and tolerability of ABM-168 monotherapy as determined by pulse rate changes from base-line in BPM (beats per minute).
Safety and tolerability-Respiratory Rate | Day 28 after last dosing.
  Safety and tolerability of ABM-168 monotherapy as determined by respiratory rate changes from base-line in breaths per minute.
Safety and tolerability-Systolic Blood Pressure | Day 28 after last dosing.
  Safety and tolerability of ABM-168 monotherapy as determined by blood pressure changes from base-line in systolic blood pressure (measured in mmHg).
Safety and tolerability-Diastolic Blood Pressure | Day 28 after last dosing.
  Safety and tolerability of ABM-168 monotherapy as determined by blood pressure changes from base-line in diastolic blood pressure (measured in mmHg).
Safety and tolerability-Ocular side effects. | Day 28 after last dosing.
  Safety and tolerability of ABM-168 monotherapy as determined by ophthalmology assessment.
Safety and tolerability-ECG parameters. | Day 28 after last dosing.
  Safety and tolerability of ABM-168 monotherapy as determined by ECGs (QT interval).
Safety and tolerability-ECOG performance | Day 28 after last dosing.
  Safety and tolerability of ABM-168 monotherapy as determined by ECOG scores (0-Fully active; - 5-Dead).
Safety and tolerability-Karnofsky performance. | Day 28 after last dosing.
  Safety and tolerability of ABM-168 monotherapy as determined by Karnofsky performance scores - 70 (able to care for self and live at home) - 100 (able to carry on normal activity).

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Indiana University Simon and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - MD Anderson Cancer Center, Houston, Texas
  - Next Oncology, Irving, Texas
  - Huntsman Cancer Institute, University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No